CLINICAL TRIAL: NCT03719937
Title: ArtificiaL Increase in chesT Wall Elastance as an alteRnative to PRONE Positioning in Moderate-to-severe ARDS: a Physiological Study The ALTERPRONE Study
Brief Title: Artificial Increase in Chest Wall Elastance as an Alternative to Prone Positioning in Moderate-to-severe ARDS.
Acronym: ALTERPRONE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Surge of COVID-19 panedemic
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Massimo Antonelli, Head of the department of Anesthesia and Intensive care medicine, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1505
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: prone positioning; chest wall mechanics; alveolar recruitment; acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: pilot-feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anterior chest wall weight (Experimental): moderate to severe ARDS patients in whom prone positioning is contraindicated. Patients will have a 100 g/kg weight placed on the anterior chest wall, while in the supine/semirecumbant position. The weights will be placed on the patients' chest for 120 minutes, and then removed. A number of measurements will be recorded before and after the procedure.
  Interventions: Device: weight on the anterior chest of the patient

INTERVENTIONS:
Device: weight on the anterior chest of the patient — The investigators aim at assessing whether and to what extent an artificial increase in chest wall elastance, while the patient is in the supine position, may yield a significant benefit to oxygenation. The increase in chest wall elastance will be will be achieved placing a 100 g/kg weight on the anterior chest wall of the patient while he/she is in the supine/semirecumbant position. The weights will be placed on the patients' chest for 120 minutes, and then removed. A number of measurements will be recorded before and after the procedure.

SUMMARY:
During moderate to severe ARDS, sessions of prone positioning lead to lung and chest wall mechanics changes that modify regional ventilation, with a final redistribution of tidal volume and PEEP towards dependent lung regions: this limits ventilator-induced lung injury, increases oxygenation and convincingly improves clinical outcome.

Physiological data indicate that the increase in chest wall elastance is crucial in determining the benefit by prone positioning on oxygenation. In some patients, however, prone positioning may not be feasible or safe due to particular comorbidities and/or technical issues.

In the present pilot-feasibility study enrolling 15 subjects with moderate to severe ARDS in whom prone positioning is contraindicated or unfeasible, we aim at assessing whether and to what extent an artificial increase in chest wall elastance while the patient is in the supine position may yield a significant benefit to oxygenation. The increase in chest wall elastance will be achieved placing 100g/kg weight on the anterior chest wall of the patient while he/she is in the supine position: this approach previoulsy appeared safe and effective in case reports and small case series. Patient's position will be standardized (30 degrees head-up, semi seated position).

This one-arm sequential study will evaluate the effects of the procedure on gas exchange, haemodynamics, lung and chest wall mechanics, alveolar recruitment (measured with the nitrogen washout-technique and multiple PV curves) and tidal volume and PEEP distribution (assessed with electrical impedance tomography).

DETAILED DESCRIPTION:
Design: Prospective, pilot, physiological study Setting: 20-bed general ICU, 13 bed surgical ICU, 10 bed neurosurgical ICU, "A. Gemelli" University hospital, Rome, Italy.

Protocol

Screening visit and oxygenation criterion validation Each patient meeting inclusion criteria will be evaluated for the presence of the oxygenation criterion. After endotracheal suctioning, eligible patients will be ventilated for 30 minutes with PEEP=5 cmH2O in the semi recumbent position and an ABG will be performed to compute PaO2/FiO2 ratio.

Patients showing PaO2/FiO2≤150 mmHg will be enrolled. Patients showing PaO2/FiO2<200 and >150 mmHg will be treated according to the standard clinical practice and reassessed for the presence of oxygenation criterion within 48 hours from the diagnosing of ARDS.

To limit the exposure to low PEEP of possibly derecruiting patient with severe oxygenation impairment, the ABG certifying the oxygenation criterion will be permitted at any time during the 30-minute monitoring period.

Procedures

All patients will be sedated, paralysed with cisatracurium infusion and connected to a ventilator equipped with lung volume measurement module (Carescape R860 - GE Healthcare, USA) through a standard bi-tube low-resistance circuit with a low-dead space, low-resistance, high-efficiency heat and moisture exchanger. For the purpose of the study, the use of heated and humidified bi-tube circuits (Fisher and Paykel healthcare, humidification chamber temperature set at 37 °C, absolute humidity provided 44 mg H2O/L) will be reserved to patients that remain hypercapnic (ph<7.30 and PaCO2>50) despite all adequate ventilator settings provided by the study protocol.

Each patient will be ventilated in volume-control mode, in the semirecumbent position (or smaller head elevation for patients with spine/pelvis movement limitations), which will not be changed throughout the study.

Ventilation settings will be standardized as follows: VT = 6 mL/Kg (predicted body weight, PBW); inspiratory flow set at 60 l/min resulting in an end-inspiratory pause of 0.2-0.5 sec, I:E ratio 1:1 to 1:3, respiratory rate tailored to achieve 45 mmHg>PaCO2>35 mmHg, PEEP set according to the clinical judgment, FiO2 set to achieve a SpO2>88-95%. A Pplat < 30 cmH2O will be considered as a safety limit.

Predicted body weight will be calculate as:

Males: PBW (kg) = 50 + 0.91 (height in cm-152) Females PBW (kg) = 45.5 + 0.91 (height in cm-152) In case of hypercapnia with Ph<7.30 despite a respiratory rate=30-35, an increase in VT up to 8 ml/kg will be allowed.

A dedicated orogastric or nasogastric tube provided with an oesophageal balloon (Cooper esophageal catheter) to monitor oesophageal pressure, estimate pleural pressure and compute transpulmonary pressure will be placed in all enrolled patients after inclusion. The adequate positioning of the esophageal catheter will be certified by an occlusion test, as previously demonstrated(15).

The GE-dedicated pneumotacograph and differential pressure transducer will be connected to the respiratory circuit to record airway pressure (PAW) and flow. The oesophageal pressure (PES) will be measured using the previously inserted oesophageal catheter, that will be connected to the auxillary pressure port of the ventilator. All the three signals will be continuously acquired by the ventilator with an analog-digital converter at a sample rate of 25 Hz (GE healthcare). A dedicated laptop connected to the ventilator will acquire PAW, PES and Flow signals through a dedicated software over the entire course of the study (Ohmeda research tool, GE healthcare).

At study enrolment, an electrical impedance tomography (EIT) belt with 16 electrodes will be placed around the thorax between the 5th or 6th parasternal intercostal space and connected to a dedicated device to record electrical impedance signals of the thorax (Swisstom EIT, Switzerland).

After included in the study, each patient will be treated as follow:

* 30-minute period in the supine position (T0);
* 120-minute period in the supine position with a 100 g/kg soft and smooth weight (warm saline bags) placed and secured on each emithorax (T1);
* 120-minute period in the supine position after the weight is removed (T2). Mechanical ventilation settings will be kept unchanged over the course of the entire study. In case of drops in the SpO2, an increase in the FiO2 will be allowed to achieve the previously described oxygenation target.

Measurements

Patient's demographics will be collected at study entry: initials, age, sex, height, weight, BMI, cause of hospital and ICU admission, SAPSII, Apache, SOFA score, date and time of ICU admission, date and time of enrolment, comorbidities, NYHA category before respiratory failure, body temperature, chest x-ray (jpeg images), chest CT scan (whether available).

During the study, each patient will undergo a standard ICU monitoring: ECG; Invasive blood pressure, SpO2, respiratory rate, diuresis.

All the relevant data follow described will be collected at prespecified timepoints.

The prespecified timepoints are:

1. baseline, T0: after the 30-minute period in the supine position (study enrolment, no weight);
2. T1a: 60 minutes after weights are positioned on the thorax;
3. T1b 120 minutes after weights are positioned on the thorax, end of T1;
4. T2a 60 minutes after weights are removed;
5. T2b 120 min after weights are removed, end of T2, end of the study;

At each timepoint the following data will be collected.

* Adverse events, if any.
* Respiratory rate, SpO2, pH, PCO2, PaO2, SaO2, PaO2/FiO2;
* Heart Rate, arterial blood pressure, central venous pressure; dosage of vasoactive or inotrope agents.
* End expiratory lung impedance (EELI) and tidal volume distribution. A ten-minute period EIT signals will be recorded and offline reviewed using a dedicated software (Swisstome EIT). Image acquisition rate will be 30 Hz. Lungs will be divided into four regions (ventral, mid-ventral, mid-dorsal and dorsal): the % of impedance variation related to tidal volume and the % EELI in the four regions as compared to the absolute values will be calculated (Appendix 3, Figures 4-5)(16).
* Respiratory mechanics End-expiratory airway pressure (PEEPAW) and the end-expiratory esophageal pressure (PEEPES) will be recorded during an 8-second expiratory hold. End-inspiratory airway pressure (PplatAW) and end-inspiratory esophageal pressure (PplatES) will be measured during a 2-second end inspiratory hold. Tidal volume (VT) will be measured as the integration of the flow-time curve during expiration.

The following parameters will be calculated offline while reviewing signals:

Airway driving pressure (∆P)=PplatAW-PEEPAW Transpulmonary end-inspiratory pressure (PplatL)=PplatAW-PplatESO Transpulmonary end-expiratory pressure (PEEPL)=PEEPAW-PEEPES Lung driving pressure (∆PL)= PplatL-PEEPL Lung plateau pressure, elastance derived (PplatL,EL)=PplatAW X (∆PL/∆P) Static respiratory system compliance (CstRS)=VT/∆P Static Lung compliance (CstL)=VT/∆PL Static Chest-wall compliance=VT/(PplatES-PEEPES) Oxygenation stretch index=PaO2/(FiO2x∆P)

• Stress and strain (measured only at T0, T1b and T2b) End-Expiratory lung volume (EELV) at the set PEEP (PEEPSET) will be measured by nitrogen washin-washout technique with a 0.2 change in the FiO2 (0.1 change in the FiO2 only allowed in case of baseline FiO2=0.9-1).

A one-breath derecruitment maneuver from PEEPSET to PEEP 0 (ZEEP) will be conducted to assess baseline functional residual capacity (FRC), that will be measured as the difference between EELV at set PEEP and the lung volume increase above FRC, measured as the difference in expired tidal volume as PEEP is decreased from 0 cmH2O in one breath with respiratory rate set at 8-10 breaths per minute. In particular, the lung volume due to the presence of set PEEP (PEEPvolume) will be measured by subtracting the insufflated VT from the expired VT (i.e. the integration of the flow signal after 5s exhalation) during a 5-second exhalation just after PEEP is reduced from set PEEP to 0.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ARDS and moderate to severe oxygenation impairment (PaO2/FiO2≤150 mmHg while receiving controlled mechanical ventilation with PEEP=5 cmH2O) will be the studied population.

   Acute respiratory failure within 1 week of a known clinical insult or new or worsening respiratory symptoms;
   * Bilateral infiltrates at the chest x-ray or CT scan, not fully explained by effusions, lobar/lung collapse, or nodules;
   * Respiratory failure not fully explained by cardiac failure or fluid overload; objective assessment required to exclude hydrostatic edema if no risk factor present.
   * PaO2/FiO2 ratio<150 mmHg after 30 mins - 1 hour of mechanical ventilation with PEEP=5 cmH2O(14).
   * Written informed consent.
2. Prone positioning deemed non-feasible by the attending clinician, or presence of at least one of the following absolute contraindications for prone positioning(5)

   * Serious facial trauma or facial surgery during the previous 15 days
   * Deep venous thrombosis treated for less than 2 days
   * Unstable spine, femur, or pelvic fractures
   * Pregnant women
   * Intracranial pressure >30 mm Hg or cerebral perfusion pressure <60 mm

Exclusion Criteria:

* Chest trauma
* Cardiothoracic surgery in the last 4/6 weeks
* Cardiac PM inserted the last 2 days
* Haemodynamic instability (MAP < 65 mmHg despite vasoactive/inotrope support)
* Chest tube with air leaks
* Presence of intrinsic PEEP > 1 cmH2O
* BMI < 18
* Height < 150 cm
* More than 48 hours from endotracheal intubation to the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
oxygenation | 120 minutes after the intervention
  PaO2/FiO2 ratio

SECONDARY OUTCOMES:
Alveolar recruitment | 1 and 2 hours after the intervention
  Changes in End expiratory lung impedance (EELI), measured with electrical impedance tomography
  A ten-minute period EIT signals will be recorded and offline reviewed using a dedicated software. Image acquisition rate will be 30 Hz. Lungs will be divided into four regions (ventral, mid-ventral, mid-dorsal and dorsal): the % of impedance variation related to tidal volume and the % EELI in the four regions as compared to the absolute values will be calculated
tidal volume dsitribution | 1 and 2 hours after the intervention
  Changes in Tidal volume distribution in 4 area of the lungs (Ventral, mid ventral, mid-dorsal, dorsal)
  A ten-minute period EIT signals will be recorded and offline reviewed using a dedicated software. Image acquisition rate will be 30 Hz. Lungs will be divided into four regions (ventral, mid-ventral, mid-dorsal and dorsal): the % of impedance variation related to tidal volume and the % EELI in the four regions as compared to the absolute values will be calculated
Lung stress | 1 and 2 hours after the intervention
  Measured at the end of an end-inspiratory occlusion, as: airway pressure - esophageal pressure + esophageal pressure at atmospheric pressure
  Static and dynamic strain will be calculated according to the following formulas:
  Lung Stress= PplatAW-PplatESO-PEEPES,ZEEP Dynamic strain = VT/FRCPEEPset Static strain= Strain due to peep ([PEEPvolume-RecZEEP at PEEP/FRCPEEPset) Pressure-volume curves at PEEP0 AND set PEEP will be conducted to confirm the reliability of the previous calculations at the end of each of the study steps
Dynamic strain | 1 and 2 hours after the intervention
  Computed as the ratio of tidal volume to functional residual capacit, with the latter measured with the nitrogen washin-washout technique
  Static and dynamic strain will be calculated according to the following formulas:
  Lung Stress= PplatAW-PplatESO-PEEPES,ZEEP Dynamic strain = VT/FRCPEEPset Static strain= Strain due to peep ([PEEPvolume-RecZEEP at PEEP/FRCPEEPset) Pressure-volume curves at PEEP0 AND set PEEP will be conducted to confirm the reliability of the previous calculations at the end of each of the study steps
Driving pressure | 1 and 2 hours after the intervention
  Respiratory system elastic pressure, measured as plateau pressure-PEEP
Transpulmonary Driving pressure | 1 and 2 hours after the intervention
  Lung elastic pressure, measured as transpulmonary plateau pressure- transpulmonary PEEP
Chest wall elastance | 1 and 2 hours after the intervention
  Elastance of abdomen/chest wall, measured as tidal change in Pes/tidal volume

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Study Chair — Catholic University of the Sacred Heart
Locations (1):
- General ICU, A. Gemelli hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Laffey JG, Bellani G, Pham T, Fan E, Madotto F, Bajwa EK, Brochard L, Clarkson K, Esteban A, Gattinoni L, van Haren F, Heunks LM, Kurahashi K, Laake JH, Larsson A, McAuley DF, McNamee L, Nin N, Qiu H, Ranieri M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators and the ESICM Trials Group. Potentially modifiable factors contributing to outcome from acute respiratory distress syndrome: the LUNG SAFE study. Intensive Care Med. 2016 Dec;42(12):1865-1876. doi: 10.1007/s00134-016-4571-5. Epub 2016 Oct 18. PMID 27757516
- [Result] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Result] Briel M, Meade M, Mercat A, Brower RG, Talmor D, Walter SD, Slutsky AS, Pullenayegum E, Zhou Q, Cook D, Brochard L, Richard JC, Lamontagne F, Bhatnagar N, Stewart TE, Guyatt G. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA. 2010 Mar 3;303(9):865-73. doi: 10.1001/jama.2010.218. PMID 20197533
- [Result] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Result] Pelosi P, Tubiolo D, Mascheroni D, Vicardi P, Crotti S, Valenza F, Gattinoni L. Effects of the prone position on respiratory mechanics and gas exchange during acute lung injury. Am J Respir Crit Care Med. 1998 Feb;157(2):387-93. doi: 10.1164/ajrccm.157.2.97-04023. PMID 9476848
- [Result] Gattinoni L, Pelosi P, Vitale G, Pesenti A, D'Andrea L, Mascheroni D. Body position changes redistribute lung computed-tomographic density in patients with acute respiratory failure. Anesthesiology. 1991 Jan;74(1):15-23. doi: 10.1097/00000542-199101000-00004. PMID 1986640
- [Result] Samanta S, Samanta S, Soni KD. Supine chest compression: alternative to prone ventilation in acute respiratory distress syndrome. Am J Emerg Med. 2014 May;32(5):489.e5-6. doi: 10.1016/j.ajem.2013.11.014. Epub 2013 Nov 13. PMID 24332252
- [Result] Mentzelopoulos SD, Roussos C, Zakynthinos SG. Prone position reduces lung stress and strain in severe acute respiratory distress syndrome. Eur Respir J. 2005 Mar;25(3):534-44. doi: 10.1183/09031936.05.00105804. PMID 15738300
- [Result] Dellamonica J, Lerolle N, Sargentini C, Beduneau G, Di Marco F, Mercat A, Richard JC, Diehl JL, Mancebo J, Rouby JJ, Lu Q, Bernardin G, Brochard L. PEEP-induced changes in lung volume in acute respiratory distress syndrome. Two methods to estimate alveolar recruitment. Intensive Care Med. 2011 Oct;37(10):1595-604. doi: 10.1007/s00134-011-2333-y. Epub 2011 Aug 25. PMID 21866369
- [Result] Ranieri VM, Giuliani R, Fiore T, Dambrosio M, Milic-Emili J. Volume-pressure curve of the respiratory system predicts effects of PEEP in ARDS: "occlusion" versus "constant flow" technique. Am J Respir Crit Care Med. 1994 Jan;149(1):19-27. doi: 10.1164/ajrccm.149.1.8111581.
- [Result] Riera J, Perez P, Cortes J, Roca O, Masclans JR, Rello J. Effect of high-flow nasal cannula and body position on end-expiratory lung volume: a cohort study using electrical impedance tomography. Respir Care. 2013 Apr;58(4):589-96. doi: 10.4187/respcare.02086. PMID 23050520
- [Result] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266
- [Result] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Result] Muders T, Luepschen H, Zinserling J, Greschus S, Fimmers R, Guenther U, Buchwald M, Grigutsch D, Leonhardt S, Putensen C, Wrigge H. Tidal recruitment assessed by electrical impedance tomography and computed tomography in a porcine model of lung injury*. Crit Care Med. 2012 Mar;40(3):903-11. doi: 10.1097/CCM.0b013e318236f452. PMID 22202705
- [Result] Pelosi P, Brazzi L, Gattinoni L. Prone position in acute respiratory distress syndrome. Eur Respir J. 2002 Oct;20(4):1017-28. doi: 10.1183/09031936.02.00401702. PMID 12412699
- [Result] Pelosi P, Cereda M, Foti G, Giacomini M, Pesenti A. Alterations of lung and chest wall mechanics in patients with acute lung injury: effects of positive end-expiratory pressure. Am J Respir Crit Care Med. 1995 Aug;152(2):531-7. doi: 10.1164/ajrccm.152.2.7633703.
- [Result] Blankman P, Hasan D, Erik G, Gommers D. Detection of 'best' positive end-expiratory pressure derived from electrical impedance tomography parameters during a decremental positive end-expiratory pressure trial. Crit Care. 2014 May 10;18(3):R95. doi: 10.1186/cc13866. PMID 24887391